CLINICAL TRIAL: NCT02856646
Title: Hodgkin Lymphoma Molecular Profiling and Clinical Outcomes in U.S. Community Oncology Practices
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-655
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Hodgkin's Disease
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population with Condition: Community Sample

SUMMARY:
The purpose of this study is to gather data on patients diagnosed with and treated for classical Hodgkin Lymphoma (cHL). It aims to closely observe how treatment for cHL is rendered, as well as assess the outcome of those treatment options and their impact on quality of life. Additional analyses will also attempt to identify prognostic or predictive biomarkers

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed diagnosis of Classical Hodgkin Lymphoma (cHL)
* Patients who are treatment-naïve, or are within ± 2 weeks beginning any line of therapy at time of enrollment
* Patients must be within ± 2 weeks of Day 1 of the first cycle of any line of therapy to enroll; a cycle is practice-defined for chemotherapy, targeted therapy, or immunotherapy-based regimens.
* Any Eastern Cooperative Oncology Group (ECOG) or Karnofsky performance status (PS)
* Patients must have available medical records for the date of diagnosis of cHL and available medical records documenting any prior treatment and treatment dates for the Hodgkin lymphoma, including chemotherapy, radiation, surgery and other anti-cancer therapy received.
* Patients must consent for use of their FFPE tissue blocks for exploratory analyses

Exclusion Criteria:

* Patients on supportive care only and not receiving anti-cancer therapy are not eligible to enroll
* Patients with unknown date of diagnosis of cHL
* Patients whose prior cHL therapy, and dates of therapy (eg, surgery, radiation, or drug therapy) are unknown
* Any other non-HL (non-Hodgkin Lymphoma) active malignancy for which the patient is receiving treatment
* Patients participating in a clinical study that does not allow enrollment into a non-interventional study
* Patients enrolled who go on to receive only supportive, palliative, hospice, or end-of-life care remain on study and should not be discontinued from follow-up.

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Composite of Treatment Patterns | Up to five years
  What are the treatment patterns of therapies used to treat cHL (ie, incorporation of novel chemotherapy or non-chemotherapy to upfront therapy, chemotherapy/radiation and/or transplant sparring patterns, incorporation of immune checkpoint agents or other investigational therapies)
Overall Survival (OS) | Up to five years
Progression Free Survival (PFS) | Up to five years
Duration of Response | Up to five years
Percentage of patients who achieve complete response | Up to 5 years
Percentage of patients who achieve partial response | Up to 5 years

SECONDARY OUTCOMES:
Health-related quality of life (HRQoL) | Up to five years
Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) | Up to five years
Drivers of Treatment Choice | Up to five years
  What are drivers of choice (eg. lack of response, safety, cost or other barriers to care) for:
  treatment decisions across and between drug classes, changes and/or discontinuation in treatment, determinants of transplant eligibility/in-eligibility?
Healthcare resource utilization measured by imputed costs | Up to five years
Grade of AE | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Norton Cancer Institute, Louisville, Kentucky, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm